CLINICAL TRIAL: NCT01581840
Title: Phase I-II on Radiochemotherapy Combined With Panitumumab in the Treatment of Localised Epidermoid Carcinoma of the Anus
Brief Title: Radiochemotherapy With Panitumumab in the Localised Epidermoid Carcinoma of the Anus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 0904
Record Dates: First submitted 2012-04-06; First posted 2012-04-20 (Estimated); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Epidermoid Carcinoma; Anus
Keywords: anus; carcinoma; panitumumab; mitomycine; 5Fu; radiotherapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — Chemoradiotherapy; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5Fu-mitomycine-panitumumab + radiotherapy (Experimental): 5 FU = 400 or 600 or 80 or 1000 mg depending of phase I results, days 1 to 4 weeks 1, 5 and 8 mitomicyne = 10 mg/m² day 1 week 1 and days 1, weeks 5 and 8 Panitumumab = 3 or 6 mg/kg (depending of phase I results) days 1, weeks: 1, 3, 5, 8 and 10
  Interventions: Drug: radiochemotherapy; Drug: Panitumumab

INTERVENTIONS:
Drug: radiochemotherapy — Radiotherapy : PTV1 45 Gy 5 weeks PTV2 20 Gy 2 weeks Chemotherapy : 5Fu (400 to 1000 mg/m²) mitomycin : 10 mg/m²
Drug: Panitumumab — 3 or 6 mg/kg (according to dose level)

SUMMARY:
Treatment is based on radiochemotherapy for locally advanced tumours. The objective of treatment is to provide a cure without resorting to abdominoperineal amputation, while preserving sphincter function.

The prognosis is mainly related to tumour size and lymph node invasion. The large majority of patients do not show any spread remote from the tumour at the time of diagnosis (2).

Recurrences are mainly of a local/regional nature and require abdominoperineal amputation. This type of intervention is not always possible or complete, which then gives rise to the particularly distressing risk of local progression, with survival at 3 years of approximately 30% (3).

It is therefore very important to achieve a complete and permanent tumour response from initial treatment with radiochemotherapy.

Furthermore, the use of an anti-EGFR antibody in combination with exclusive radiotherapy in ENT cancer was able to increase recurrence-free survival and overall survival in these patients. These data are in favour of the use of a combination of chemotherapy and anti-EGFR antibodies in epidermoid cancer of the anus.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven epidermoid carcinoma of the anus
* Locally advanced tumour without metastases
* Stage T2>3 cm or T3 or T4, irrespective of N
* Stage N1-N3 irrespective of T stage (T1 to T4)
* General condition WHO 0-1
* Life expectancy > 3 months
* Signed informed consent form
* Age > 18 years
* Effective contraception in female and/or male patients having reached sexual maturity during treatment and up to 6 months after the end of treatment
* CD4 > 400 / mm3
* Measureable tumor on at least one of the following exams : MRI, endoscopic ultrasonography, clinical exam

Exclusion Criteria:

* Presence of metastases
* Previous anti-EGFR therapy
* Stage T1N0 or T2 < 3 cm N0
* History of pelvic radiotherapy
* At least one of the following laboratory test results: Neutrophils < 1500 /mm3, platelets < 100 000 /mm3, Hb < 9 g/dl, leukocytes < 3000/mm3, blood bilirubin > 1.5 times the upper limit of the normal range, transaminase (ASAT and ALAT) > 2.5 times the upper limit of the normal range, creatinine clearance < 50 mL/min (Cockcroft's formula Appendix x), Mg2+ < the lower limit of the normal range, Ca2+ < the lower limit of the normal range
* Significant coronary artery disease or myocardial infarction in the past year
* Follow-up not possible due to psychological or geographic reasons
* History of interstitial pneumonitis or pulmonary fibrosis
* History of malignant disease in the past five years apart from basocellular skin carcinoma or in situ cervical carcinoma having received adequate treatment
* Pregnant or breast-feeding women, women of child-bearing potential not having taken a pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique VENDRELY, MD, Principal Investigator — Hôpital Haut-Lévêque - Bordeaux
Locations (15):
- France (15):
  - Pessac - Hôpital Haut Lévêque, Bordeaux
  - CH - Hopitaux civils de Colmar, Colmar
  - Centre d'oncologie et de radiothérapie du Parc, Dijon
  - Centre Oscar Lambret, Lille
  - CH - CHBS - Hôpital du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Régional du Cancer Montpellier, Montpellier
  - Clinique Privée - Plein Ciel, Mougins
  - Institut Curie, Paris
  - Cario - HPCA - Hôpital privé des Côtes D'Armor, Plérin
  - CH - Annecy Genevois, Pringy
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud
  - CHU, Saint-Priest-en-Jarez
  - CAC - Paul Strauss, Strasbourg

REFERENCES:
- [Result] Vendrely V, Lemanski C, Gnep K, Barbier E, Hajbi FE, Lledo G, Dahan L, Terrebonne E, Manfredi S, Mirabel X, Mammar V, Cowen D, Lepage C, Aparicio T; for FFCD investigators/Collaborators. Anti-epidermal growth factor receptor therapy in combination with chemoradiotherapy for the treatment of locally advanced anal canal carcinoma: Results of a phase I dose-escalation study with panitumumab (FFCD 0904). Radiother Oncol. 2019 Nov;140:84-89. doi: 10.1016/j.radonc.2019.05.018. Epub 2019 Jun 8. PMID 31185328
- [Derived] Vendrely V, Ronchin P, Minsat M, Le Malicot K, Lemanski C, Mirabel X, Etienne PL, Lievre A, Darut-Jouve A, de la Fouchardiere C, Giraud N, Breysacher G, Argo-Leignel D, Thimonnier E, Magne N, Abdelghani MB, Lepage C, Aparicio T; for FFCD investigators/Collaborators. Panitumumab in combination with chemoradiotherapy for the treatment of locally-advanced anal canal carcinoma: Results of the FFCD 0904 phase II trial. Radiother Oncol. 2023 Sep;186:109742. doi: 10.1016/j.radonc.2023.109742. Epub 2023 Jun 12. PMID 37315583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2016 and November 2017 (Phase II), 45 patients were enrolled by 15 french centers
Groups:
- 5Fu-mitomycine-panitumumab + Radiotherapy: 5 FU = 400 mg days 1 to 4 weeks 1, 5 and 8 mitomicyne = 10 mg/m² day 1 week 1 and days 1, weeks 5 and 8 Panitumumab = 3 mg/kg days 1, weeks: 1, 3, 5, 8 and 10
  radiochemotherapy: Radiotherapy : PTV1 45 Gy 5 weeks PTV2 20 Gy 2 weeks
Period: Overall Study
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.19 [56.50 to 67.20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 45
Region of Enrollment [Number; unit: participants]
  France | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Response to Treatment
Description: Complete response was defined by the complete disappearance of the tumor on proctological examination and morphological examinations (MRI and/or echo-endoscopy) and the absence of secondary lesion appearance. The responses were validated by an independent committee:
  * In the event of a discrepancy between the investigator and the independent committee, the independent committee's response was used;
  * in case of uncertainty of the investigator on the response, the committee decided on the response in view of the clinical and morphological data; This endpoint was assessed 8 weeks after the end of treatment (week 15). A patient who died (regardless of cause) was considered a failure for the primary endpoint
Time Frame: 8 weeks evaluations after the end of the treatment by radiochemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
Number analyzed (Participants) | 45
Participants
  Complete response | 30
  Partial response | 10
  Stability | 0
  Progression | 4
  Death before the evaluation | 1

2. Secondary Outcome: Percentage of Patients With Complete Response to Treatment
Description: Complete response was defined by the complete disappearance of the tumor on proctological examination and morphological examinations (MRI and/or echo-endoscopy) and the absence of secondary lesion appearance according to the investigator's opinion
Time Frame: 16 weeks after the end of the treatement by radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
Number analyzed (Participants) | 44
Participants
  Complete response | 27
  Partial response | 9
  Stability | 1
  Progression | 7

3. Secondary Outcome: 3 Years Colostomy-free Survival (CFS)
Description: It was defined as the time from inclusion to the date of colostomy or death (from any cause). Patients alive without colostomy were censored at date of last news. If a patient had a shunt colostomy and continuity wasrestored, the patient was counted among the patients without a colostomy.
Time Frame: At 3 years after inclusion
Measure: Number (95% Confidence Interval); unit: % of patients Colostomy-free at 3 years
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
Number analyzed (Participants) | 45
% of patients Colostomy-free at 3 years | 68.8 [53.1 to 80.2]

4. Secondary Outcome: Recurrence-free Survival (RFS) at 3 Years
Description: It was defined as the time from inclusion to the date of first recurrence (local, regional, metastatic and second anal cancer) or death. Patients alive without recurrence were censored at date of last news.
Time Frame: At 3 years after inclusion
Measure: Number (95% Confidence Interval); unit: % of pts with Reccurence-free at 3 yrs
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
Number analyzed (Participants) | 45
% of pts with Reccurence-free at 3 yrs | 62.2 [46.5 to 74.6]

5. Secondary Outcome: Overall Survival (OS) at 12 Months
Description: The percentage was evaluated at 12 months using the Kaplan Meier estimation.
  In the safety part all the death collected during the study will be reported.
Time Frame: At 12 months after inclusion
Measure: Number (95% Confidence Interval); unit: % of patients alive at 12 months
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
Number analyzed (Participants) | 45
% of patients alive at 12 months | 95.6 [83.5 to 99.7]

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 3 years after start of treatment Adverse Events were assessed up to 12 months
Arm/Group | 5Fu-mitomycine-panitumumab + Radiotherapy
All-Cause Mortality (participants affected / at risk) | 10/45
Serious Adverse Events (participants affected / at risk) | 14/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5Fu-mitomycine-panitumumab + Radiotherapy (N=45)
Vaginal fistula (Reproductive system and breast disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 1
Small bowel inflamation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small bowel obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Cutaneous infection (Infections and infestations) | 1
Septicemia (Infections and infestations) | 1
Lymphocytes decreased (Investigations) | 1
Complication of vascular access (Injury, poisoning and procedural complications) | 1
Hypokaliemia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5Fu-mitomycine-panitumumab + Radiotherapy (N=45)
Erythema (Skin and subcutaneous tissue disorders) | 25
Prurit (Skin and subcutaneous tissue disorders) | 12
Acneiform rash (Skin and subcutaneous tissue disorders) | 25
Cutaneous rash (Skin and subcutaneous tissue disorders) | 11
Vulvar and vaginal inflammation (Reproductive system and breast disorders) | 22
Cystitis (Renal and urinary disorders) | 19
Pollakiurie (Renal and urinary disorders) | 7
Diarrhea (Gastrointestinal disorders) | 34
Abdominal pain (Gastrointestinal disorders) | 10
Anal pain (Gastrointestinal disorders) | 19
Mucositis (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 24
Proctitis/Rectitis (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 12
Anemia (Blood and lymphatic system disorders) | 30
Radiation Dermatitis (Injury, poisoning and procedural complications) | 14
Anorexia (Metabolism and nutrition disorders) | 29
Hypokaliemia (Metabolism and nutrition disorders) | 9
Fatigue (General disorders) | 35
Fever (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT01581840/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT01581840/SAP_001.pdf